CLINICAL TRIAL: NCT06689462
Title: Appraisal of the Modified Cancer Cachexia Index in Locally Advanced Gastric Cancer Patients Undergoing Neoadjuvant Chemotherapy
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Other Study IDs: 2024NLAGCCachexia; 2022QNA026 (Other Grant/Funding Number: Chang-Ming Huang)
Record Dates: First submitted 2024-11-13; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer; Neoadjuvant Chemotherapy; Computed Tomography; Random Forest Model
Keywords: Cancer cachexia index; Locally Advanced Gastric Cancer; Neoadjuvant chemotherapy; Adjuvant chemotherapy; Survival
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this study, consecutive 600 patients with LAGC(cT2-4NanyM0) who underwent NACT between Jan. 2010 and Jun. 2022 were identified from two tertiary hospitals. The mCXI was constructed based on Random Forest model, calculated as (post-NACT L3 subcutaneous adipose tissue area [SAT])×(post-NACT serum albumin [ALB])/(post-NACT platelet count [PLT]). Patients were categorized into two subgroups: mCXI-low and mCXI-high. mCXI is associated with the overall prognosis in patients with locally advanced gastric cancer underwent neoadjuvant chemotherapy, is superior to traditional CXI, and may serve as a decision-making tool for guiding personalized postoperative adjuvant chemotherapy.

DETAILED DESCRIPTION:
This is a multicenter retrospective cohort study

ELIGIBILITY:
Inclusion Criteria:

* (1) locally advanced gastric cancer (cT2-4NxM0) with clinical staging before neoadjuvant chemotherapy, (2) no history of other malignant tumors, (3) no evidence of distant metastasis or invasion of adjacent organs, and (4) patients who underwent radical gastrectomy following neoadjuvant chemotherapy.

Exclusion Criteria:

* (1) history of gastric surgery; (2) acute cardiovascular disease (such as cerebrovascular or coronary artery injury) within the past three months; (3) emergency surgery; (4) active infection or severe systemic immunodeficiency; and (5) incomplete serological, computed tomography, or anthropometric data.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with locally advanced gastric cancer (cT2-4NanyM0)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-13 (Actual)

PRIMARY OUTCOMES:
3-year overall survival | 3 years or 36 months.
  Survival status at 3 years: survival, death, the end of surgery to death.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, M.D. FACS, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No